CLINICAL TRIAL: NCT04999839
Title: A Phase 2b, Randomized, Multicenter, Double-blind, Placebo-controlled, Multiple-dose Study to Evaluate the Efficacy, Safety, and Tolerability of NDI-034858 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Study of NDI-034858 in Participants With Moderate to Severe Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Innovaderm Research Inc. (Other); Nimbus Lakshmi, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4858-201
Record Dates: First submitted 2021-07-19; First posted 2021-08-11 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Moderate to Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo matched to NDI-034858 oral capsules, once daily (QD) for up to 12 weeks.
  Interventions: Other: Placebo
- NDI-034858 2 milligrams (mg) (Experimental): Participants received 2 mg of NDI-034858 oral capsules, QD for up to 12 weeks.
  Interventions: Drug: NDI-034858 study drug
- NDI-034858 5 mg (Experimental): Participants received 5 mg of NDI-034858 oral capsules, QD for up to 12 weeks.
  Interventions: Drug: NDI-034858 study drug
- NDI-034858 15 mg (Experimental): Participants received 15 mg of NDI-034858 oral capsules, QD for up to 12 weeks.
  Interventions: Drug: NDI-034858 study drug
- NDI-034858 30 mg (Experimental): Participants received 30 mg (2*15 mg) of NDI-034858 oral capsules, QD for up to 12 weeks.
  Interventions: Drug: NDI-034858 study drug

INTERVENTIONS:
Drug: NDI-034858 study drug — NDI-034858 2 mg oral capsules.
  Other Names: NDI-034858; TAK-279
  Arms: NDI-034858 2 milligrams (mg)
Drug: NDI-034858 study drug — NDI-034858 5 mg oral capsules.
  Other Names: NDI-034858; TAK-279
  Arms: NDI-034858 5 mg
Drug: NDI-034858 study drug — NDI-034858 15 mg oral capsules.
  Other Names: NDI-034858; TAK-279
  Arms: NDI-034858 15 mg
Drug: NDI-034858 study drug — NDI-034858 30 mg (2*15 mg) oral capsules.
  Other Names: NDI-034858; TAK-279
  Arms: NDI-034858 30 mg
Other: Placebo — Placebo matched to NDI-034858 oral capsules.
  Other Names: Non Active Ingredient
  Arms: Placebo

SUMMARY:
This is a Phase 2b, randomized, multicenter, double-blind, placebo-controlled, multiple-dose study designed to evaluate the efficacy, safety, and tolerability of NDI-034858 in participants with moderate to severe plaque psoriasis. This study will also evaluate the plasma concentrations of NDI-034858 and explore the immune response to NDI-034858 in participants with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
Approximately 259 male and female participants, aged 18 to 70 years (inclusive) were enrolled in this study. Participants were randomized to receive either one of the four doses of NDI-034858, or placebo on Day 1. The goal was to have approximately 50 participants randomized per treatment group (1:1:1:1:1 ratio) on Day 1. During the treatment period, NDI-034858 or placebo was orally administered QD for 12 weeks. The 12 week treatment period was followed by a 4-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a participant must meet all of the following criteria, either at the screening and Day 1 visits or only at one of the specified visits (screening or Day 1) as noted in the criterion:

1. Male or female participant aged 18 to 70 years, inclusive, at the time of consent.
2. Participant has a history of plaque psoriasis for at least 6 months prior to the screening visit.
3. Participant had no significant flare in psoriasis for at least 3 months before screening (information obtained from medical chart or participant's physician, or directly from the participant).
4. Participant has moderate to severe plaque psoriasis as defined by a PASI score ≥ 12 and a PGA score ≥ 3 at screening and Day 1.
5. Participant has plaque psoriasis covering ≥ 10% of his or her total BSA at screening and Day 1.
6. Participant must be a candidate for phototherapy or systemic therapy.
7. For female participants of childbearing potential involved in any sexual intercourse that could lead to pregnancy: the participant must agree to use a highly effective contraceptive method from at least 4 weeks prior to Day 1 until at least 4 weeks after the last study product administration. Highly effective contraceptive methods include hormonal contraceptives (eg, combined oral contraceptive, patch, vaginal ring, injectable, or implant), intrauterine devices or intrauterine systems, vasectomized partner(s) (provided vasectomy was performed ≥ 4 months prior to screening), bilateral tubal ligation or occlusion, or double barrier methods of contraception (eg, male condom with cervical cap, male condom with diaphragm, and male condom with contraceptive sponge) in conjunction with spermicide.
8. Female participants of childbearing potential have had a negative serum pregnancy test at screening and negative urine pregnancy test at Day 1.
9. For male participants involved in any sexual intercourse that could lead to pregnancy, participant must agree to use one of the highly effective contraceptive methods listed in Inclusion Criterion 6, from Day 1 until at least 12 weeks after the last study product administration. If the female partner of a male participant uses any of the hormonal contraceptive methods listed above, this contraceptive method should be used by the female partner from at least 4 weeks before Day 1 until at least 12 weeks after the last study product administration.
10. Participant has a BMI within the range of 18 to 42 kg/m2, inclusive (BMI = weight [kg]/[height (m)]2), and total body weight >50 kg (110 lb).
11. Participant is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
12. Participant must be willing to comply with all study procedures and must be available for the duration of the study.

Exclusion Criteria:

A participant who meets any of the following criteria at the screening and/or Day 1 visits, as applicable, will be excluded from participation in this study:

1. Participant is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study.
2. Participant has evidence of erythrodermic, pustular, predominantly guttate psoriasis, or drug induced psoriasis.
3. Participant has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
4. Participant has immune-mediated conditions commonly associated with psoriasis, such as psoriatic arthritis, uveitis, inflammatory bowel disease, that require systemic treatment (including corticosteroids, immunosuppressants, or biologics). Note: Participants with immune-mediated conditions that do not require systemic treatment may be included in the study. Certain therapies such as NSAIDs may be permitted, but should be discussed with the Medical Monitor prior to determination of participant eligibility.
5. Participant has any clinically significant medical condition, evidence of an unstable clinical condition (eg, cardiovascular, renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, immunologic, or local active infection/infectious illness), psychiatric condition, or vital signs/physical/laboratory/ECG abnormality that would, in the opinion of the investigator, put the participant at undue risk or interfere with interpretation of study results.
6. Participant had a major surgery within 8 weeks prior to Day 1 or has a major surgery planned during the study.
7. Participant has a history of Class III or IV congestive heart failure as defined by New York Heart Association Criteria.
8. Participant has been hospitalized in the past 3 months for asthma, has ever required intubation for treatment of asthma, currently require oral corticosteroids for the treatment of asthma, or has required more than one short-term (≤ 2 weeks) course of oral corticosteroids for asthma within 6 months prior to Day 1.
9. Participant has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Participant with successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded.
10. Participant has a history of fever, inflammation, or systemic signs of illness suggestive of systemic or invasive infection within 4 weeks prior to Day 1.
11. Participant has an active bacterial, viral, fungal, mycobacterial infection, or other infection (including TB or atypical mycobacterial disease), or any major episode of infection that required hospitalization or treatment with intravenous antibiotics within 12 weeks prior to Day 1, or oral antibiotics within 4 weeks prior to Day 1.
12. Participant has a history of chronic or recurrent infectious disease, including but not limited to chronic renal infection, chronic chest infection, recurrent urinary tract infection, fungal infection (with the exception of superficial fungal infection of the nailbed), or infected skin wounds or ulcers.
13. Participant has a history of an infected joint prosthesis or has received antibiotics for a suspected infection of a joint prosthesis, if that prosthesis has not been removed or replaced.
14. Participant has active herpes infection, including herpes simplex 1 and 2 and herpes zoster (demonstrated on physical examination and/or medical history) within 8 weeks prior to Day 1.
15. Participant has a history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status in the opinion of the investigator (eg, history of splenectomy, primary immunodeficiency).
16. Participant has positive results for hepatitis B surface antigens (HBsAg), antibodies to hepatitis B core antigens (anti-HBc), hepatitis C virus (HCV), or human immunodeficiency virus (HIV).
17. Participant has clinical or laboratory evidence of active or latent TB infection at screening.
18. Participant with any of the following laboratory values at the screening visit:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values ≥ 3 times the upper limit of normal (ULN);
    2. Hemoglobin < 11.0 g/dL (< 110.0 g/L);
    3. White blood cell count < 3.5 x 109/L (< 3500/mm3);
    4. Absolute neutrophil count of < 1.8 x 109/L (< 1800/mm3);
    5. Absolute lymphocyte count of < 1.0 x 109/L (< 1000/mm3);
    6. Platelet count < 100 x 109/L (< 100,000/mm3);
    7. Total bilirubin ˃ 2 times the ULN.
19. Participant who have given > 50 ml of blood or plasma within 30 days of screening or > 500 mL of blood or plasma within 56 days of screening (during a clinical study or at a blood bank donation).
20. Participant has used any topical medication that could affect psoriasis (including corticosteroids, retinoids, vitamin D analogues [such as calcipotriol], JAK inhibitors, or tar) within 2 weeks prior to Day 1.
21. Participant has used any systemic treatment that could affect psoriasis (including oral, intravenous, intraarticular, intrathecal, intramuscular, or intralesional corticosteroids, oral retinoids, immunosuppressive/immunomodulating medication, methotrexate, cyclosporine, oral JAK inhibitors, or apremilast) within 4 weeks prior to Day 1.
22. Participant has received any UV-B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to Day 1.
23. Participant has had PUVA treatment within 4 weeks prior to Day 1.
24. Participant has received any live-attenuated vaccine within 4 weeks prior to Day 1 or plans to receive a live-attenuated vaccine during the study and up to 4 weeks or 5 half lives of the study product, whichever is longer, after the last study product administration. Note: Nonlive-attenuated vaccines or boosters for Coronavirus Disease 2019 (COVID-19) (eg, RNA-based vaccines, inactivated adenovirus-based vaccines, protein-based vaccines) are allowed during the study. The study site should follow local guidelines related to COVID-19.
25. Participant is currently receiving a nonbiological investigational product or device or has received one within 4 weeks prior to Day 1.
26. Participant has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1 (except those listed in Exclusion Criterion 27 and 28 that are to be excluded for 6 months).
27. Participant was previously enrolled in any study with NDI-034858.
28. Participant has a history of lack of response to any therapeutic agent targeting IL-12, IL-17, and/or IL 23 (eg, ustekinumab, secukinumab, ixekizumab, brodalumab, guselkumab, tildrakizumab, risankizumab) at approved doses after at least 12 weeks of therapy, and/or received one of these therapies within 6 months prior to Day 1.
29. Participant has received rituximab or other immune-cell depleting therapy within 6 months.
30. Participant is currently being treated with strong or moderate cytochrome P450 3A (CYP3A4) inhibitors (such as itraconazole), or has received moderate or strong CYP3A4 inhibitors within 4 weeks prior to Day 1.
31. Participant is currently being treated with terbinafine, or has received terbinafine within 4 weeks prior to Day 1.
32. Participant has consumed grapefruit within 1 week prior to Day 1.
33. Participant has used tanning booths within 4 weeks prior to Day 1, has had excessive sun exposure, or is not willing to minimize natural and artificial sunlight exposure during the study.
34. Participant has a known or suspected allergy to NDI-034858 or any component of the investigational product, or any other significant drug allergy (such as anaphylaxis or hepatotoxicity).
35. Participant has a known history of clinically significant drug or alcohol abuse in the last year prior to Day 1.
36. For participant consenting to biopsy collection only:

    * Participant has a history of an allergic reaction or significant sensitivity to lidocaine or other local anesthetics.
    * Participant has a history of hypertrophic scarring or keloid formation in scars or suture sites.
    * Participant has taken anticoagulant medication, such as heparin, low molecular weight (LMW)-heparin, warfarin, or antiplatelet agents (except low-dose aspirin ≤ 81 mg which will be allowed), within 2 weeks prior to Day 1, or has a contraindication to skin biopsies. Nonsteroidal anti-inflammatory drugs will not be considered antiplatelet agents and will be allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (69):
- United States (59):
  - Nimbus site 137, Birmingham, Alabama
  - Nimbus site 156, Birmingham, Alabama
  - Nimbus site 132, Scottsdale, Arizona
  - Nimbus site 133, Bryant, Arkansas
  - Nimbus site 134, Fountain Valley, California
  - Nimbus site 108, Los Angeles, California
  - Nimbus site 124, Sacramento, California
  - Nimbus site 153, San Diego, California
  - Nimbus site 111, San Diego, California
  - Nimbus site 148, Santa Rosa, California
  - Nimbus site 120, Sherman Oaks, California
  - Nimbus site 155, Doral, Florida
  - Nimbus site 149, Hialeah, Florida
  - Nimbus site 130, Largo, Florida
  - Nimbus site 160, Margate, Florida
  - Nimbus site 107, Miami Lakes, Florida
  - Nimbus site 139, Miami Lakes, Florida
  - Nimbus site 118, Ocala, Florida
  - Nimbus site 157, Sweetwater, Florida
  - Nimbus site 101, Tampa, Florida
  - Nimbus site 102, Tampa, Florida
  - Nimbus site 116, West Palm Beach, Florida
  - Nimbus site 147, Columbus, Georgia
  - Nimbus site 150, Macon, Georgia
  - Nimbus site 119, Sandy Springs, Georgia
  - Nimbus site 123, Skokie, Illinois
  - Nimbus site 159, Clarksville, Indiana
  - Nimbus site 140, Indianapolis, Indiana
  - Nimbus site 154, Overland Park, Kansas
  - Nimbus site 161, Louisville, Kentucky
  - Nimbus site 105, Louisville, Kentucky
  - Nimbus site 136, Lake Charles, Louisiana
  - Numbus site 114, Metairie, Louisiana
  - Nimbus site 122, Rockville, Maryland
  - Nimbus site 115, Beverly, Massachusetts
  - Nimbus site 135, Quincy, Massachusetts
  - Nimbus site 146, Ann Arbor, Michigan
  - Nimbus site 103, Bay City, Michigan
  - Nimbus site 112, Troy, Michigan
  - Nimbus site 138, Troy, Michigan
  - Nimbus site 158, New Brighton, Minnesota
  - Nimbus site 143, New York, New York
  - Nimbus site 129, Charlotte, North Carolina
  - Nimbus site 106, Wilmington, North Carolina
  - Nimbus site 127, Bexley, Ohio
  - Nimbus site 145, Columbus, Ohio
  - Nimbus site 128, Fairborn, Ohio
  - Nimbus site 141, Norman, Oklahoma
  - Nimbus site 125, Pittsburgh, Pennsylvania
  - Nimbus site 110, Charleston, South Carolina
  - Nimbus site 117, Jackson, Tennessee
  - Nimbus site 121, Nashville, Tennessee
  - Nimbus site 109, Arlington, Texas
  - Nimbus site 113, Bellaire, Texas
  - Nimbus site 131, Katy, Texas
  - Nimbus site 104, San Antonio, Texas
  - Nimbus site 152, San Antonio, Texas
  - Nimbus site 162, Webster, Texas
  - Nimbus site 142, Spokane, Washington
- Canada (10):
  - Nimbus site 204, Calgary
  - Nimbus site 206, Calgary
  - Nimbus site 212, Edmonton
  - Nimbus site 209, Hamilton
  - Nimbus site 203, Markham
  - Nimbus site 201, Montreal
  - Nimbus site 205, Oshawa
  - Nimbus site 210, Peterborough
  - Nimbus site 208, Red Deer
  - Nimbus site 202, Waterloo

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Armstrong AW, Gooderham M, Lynde C, Maari C, Forman S, Green L, Laquer V, Zhang X, Franchimont N, Gangolli EA, Blau J, Zhao Y, Zhang W, Srivastava B, Heap G, Papp K. Tyrosine Kinase 2 Inhibition With Zasocitinib (TAK-279) in Psoriasis: A Randomized Clinical Trial. JAMA Dermatol. 2024 Oct 1;160(10):1066-1074. doi: 10.1001/jamadermatol.2024.2701. PMID 39167366
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/4b255e32353e400a

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 55 study centers in the United States and Canada from 11 August 2021 to 12 September 2022.
Pre-assignment Details: A total of 259 participants received either one of the four doses of NDI-034858 (2 milligrams [mg], 5 mg, 15 mg, or 30 mg), or matching placebo.
Groups:
- NDI-034858 2 mg: Participants received 2 mg of NDI-034858 oral capsules, QD for up to 12 weeks.
Period: Overall Study
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Started | 52 | 50 | 52 | 53 | 52
Completed | 43 | 42 | 45 | 46 | 47
Not Completed | 9 | 8 | 7 | 7 | 5
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2 | 4 | 1
Not completed — Withdrawal by Subject | 6 | 5 | 3 | 2 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor request | 0 | 1 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The modified intent-to-treat (mITT) analysis set included all participants who were randomized and received at least one dose of study treatment.
Groups:
- Placebo: Participants received placebo matched to NDI-034858 oral capsules, QD for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg | Total
Number analyzed (Participants) | 52 | 50 | 52 | 53 | 52 | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.70) | 45.8 (14.17) | 45.1 (13.60) | 46.2 (13.02) | 48.5 (11.41) | 46.9 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 11 | 19 | 19 | 82
  Male | 31 | 38 | 41 | 34 | 33 | 177
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 21 | 12 | 19 | 15 | 93
  Not Hispanic or Latino | 26 | 29 | 40 | 34 | 37 | 166
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 2 | 5
  Asian | 5 | 3 | 7 | 2 | 3 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 4 | 3 | 4 | 17
  White | 44 | 43 | 40 | 46 | 42 | 215
  More than one race | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Psoriasis Area and Severity Index (PASI) [Mean (Standard Deviation); unit: score on a scale] — PASI quantifies severity of a participant's psoriasis based on both "lesion severity" and "percent of BSA" affected. PASI: composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk, and lower limbs) with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. PASI composite score varies in increments of 0.1 and range from 0 (no disease) to 72 (maximal disease), with higher scores = greater severity of psoriasis.
  score on a scale | 18.27 (8.120) | 18.37 (6.752) | 18.60 (6.050) | 15.52 (4.504) | 17.63 (6.220) | 17.67 (6.477)
Dermatology Life Quality Index (DLQI) [Mean (Standard Deviation); unit: score on a scale] — The DLQI is a simple 10 question validated questionnaire that has been used in more than 40 different skin conditions. It is the most frequently used quality of life instrument in studies of randomized controlled trials in dermatology. Each question is scored on a four-point Likert scale: very much (3); a lot (2); a little (1); not at all (0). DLQI total score is defined as the sum of the 10 questions, ranging from 0 (not at all) to 30 (very much). Higher scores indicate more impact on quality of life of participants; and lower scores indicate less impact on quality of life of participants.
  score on a scale | 12.4 (7.04) | 10.3 (6.19) | 12.8 (7.45) | 11.9 (7.10) | 12.5 (6.87) | 12.0 (6.95)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved at Least 75 Percent (%) Improvement From Baseline in Psoriasis Area and Severity Index (PASI-75) at Week 12
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of body surface area (BSA)" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI composite score varies in increments of 0.1 and range from 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. PASI 75 response is a binary measure defined as at least a 75% improvement in PASI score at Week 12, relative to baseline PASI score.
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all participants who were randomized and received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 52 | 50 | 52 | 53 | 52
percentage of participants | 5.8 | 18.0 | 44.2 | 67.9 | 67.3
Statistical Analysis 1: Comparison: Placebo vs NDI-034858 2 mg; Test type: Superiority; p = 0.052, Cochran-Mantel-Haenszel — P-value was calculated using a Cochran-Mantel-Haenszel (CMH) test, with prior treatment with biologics included as a stratification factor, comparing the percentage of participants in each dose of NDI-034858 vs placebo; Odds Ratio (OR) = 3.727, 95% CI 2-sided [0.933 to 14.885] — Odds ratio for achievement of PASI-75 was calculated using the Mantel-Haenszel (MH) method
Statistical Analysis 2: Comparison: Placebo vs NDI-034858 5 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — P-value was calculated using a CMH test, with prior treatment with biologics included as a stratification factor, comparing the percentage of participants in each dose of NDI-034858 vs placebo; Odds Ratio (OR) = 12.733, 95% CI 2-sided [3.525 to 45.994] — Odds ratio for achievement of PASI-75 was calculated using the MH method
Statistical Analysis 3: Comparison: Placebo vs NDI-034858 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 29.014, 95% CI 2-sided [8.526 to 98.735] — Odds ratio for achievement of PASI-75 was calculated using the MH method
Statistical Analysis 4: Comparison: Placebo vs NDI-034858 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 2]; Odds Ratio (OR) = 40.111, 95% CI 2-sided [10.277 to 156.548] — Odds ratio for achievement of PASI-75 was calculated using the MH method

2. Secondary Outcome: Percentage of Participants Who Achieved Physician's Global Assessment (PGA) Score of Clear (0) or Almost Clear (1) at Week 12
Description: The PGA is a global assessment of the current state of the disease. It is a 5-point morphological assessment of overall disease severity with scores ranging from 0 to 4, where Score 0: Clear (No signs of psoriasis; post-inflammatory hyperpigmentation may be present); Score 1: Almost clear (No thickening; normal to pink coloration; no to minimal focal scaling); Score 2: Mild (Just detectable to mild thickening; pink to light red coloration; predominantly fine scaling); Score 3: Moderate (Clearly distinguishable to moderate thickening; dull to bright red; clearly distinguishable to moderate erythema; moderate scaling); Score 4: Severe (Severe thickening with hard edges; bright to deep dark red coloration; severe/coarse scaling covering almost all or all lesions). The percentage of participants who achieved a PGA score of clear (0) or almost clear (1) at Week 12 were reported.
Time Frame: At Week 12
Population: The mITT analysis set included all participants who were randomized and received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 52 | 50 | 52 | 53 | 52
percentage of participants | 3.8 | 10.0 | 26.9 | 49.1 | 51.9

3. Secondary Outcome: Percentage of Participants Who Achieved at Least 90% Improvement From Baseline in Psoriasis Area and Severity Index (PASI-90) at Week 12
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI composite score varies in increments of 0.1 and range from 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. PASI 90 response is a binary measure defined as at least a 90% improvement in PASI score at Week 12, relative to baseline PASI score.
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all participants who were randomized and received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 52 | 50 | 52 | 53 | 52
percentage of participants | 0 | 8.0 | 21.2 | 45.3 | 46.2

4. Secondary Outcome: Percentage of Participants Who Achieved at Least 100% Improvement From Baseline in Psoriasis Area and Severity Index (PASI-100) at Week 12
Description: The PASI quantifies the severity of a participant's psoriasis based on both "lesion severity" and the "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI composite score varies in increments of 0.1 and range from 0 (no disease) to 72 (maximal disease), with higher scores representing greater severity of psoriasis. PASI 100 response is a binary measure defined as at least a 100% improvement in PASI score at Week 12, relative to baseline PASI score.
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all participants who were randomized and received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 52 | 50 | 52 | 53 | 52
percentage of participants | 0 | 2.0 | 9.6 | 15.1 | 32.7

5. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score at Week 12
Description: The DLQI is a simple 10 question validated questionnaire that has been used in more than 40 different skin conditions. The DLQI is the most frequently used quality of life instrument in studies of randomized controlled trials in dermatology. Each question is scored on a four-point Likert scale: very much (3); a lot (2); a little (1); not at all (0). DLQI total score is defined as the sum of the 10 questions, ranging from 0 (not at all) to 30 (very much). Higher scores indicate more impact on quality of life of participants; and lower scores indicate less impact on the quality of life of participants.
Time Frame: Baseline, Week 12
Population: The mITT analysis set included all participants who were randomized and received at least one dose of study treatment. Overall number of participants analyzed signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 47 | 43 | 47 | 46 | 47
score on a scale | -4.9 (0.75) | -5.3 (0.78) | -7.9 (0.75) | -8.5 (0.74) | -8.9 (0.75)

6. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Event (TEAEs) and Serious TEAEs
Description: An adverse event (AE) means any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product whether or not it is related to the medicinal product. TEAEs were defined as any AEs with onset date on or after the first study treatment dosing. An SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality or birth defect, an important medical event. TEAEs included both serious and non-serious AEs.
Time Frame: From start of study drug administration up to Week 16
Population: The safety analysis set included all participants who received at least one dose of the study product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 52 | 50 | 52 | 53 | 52
Participants
  Participants with TEAEs | 23 | 31 | 28 | 28 | 31
  Participants with Serious TEAEs | 0 | 0 | 0 | 1 | 0

7. Secondary Outcome: Plasma Concentrations of NDI-034858 in Participants Receiving Active Treatment
Description: The analysis of NDI-034858 levels in plasma was performed using a validated reversed-phase Ultra High-Performance Liquid Chromatography coupled with tandem mass-spectrometry (UHPLC-MS/MS) method. Here, plasma concentrations of NDI-034858 determined at given timepoints were reported.
Time Frame: Week 1: Day 1, Pre-dose and 1-hour post-dose; Week 4: Pre-dose, 1-hour and 4 hours post-dose; Week 8: Pre-dose; Week 12: Post-dose
Population: The pharmacokinetic (PK) analysis set included all participants who received at least one dose of NDI-034858 and had evaluable plasma concentration data. One participant had PK data missing at baseline (Week 1, Day 1: pre-dose) in 30 mg arm but contributed to PK analysis at post baseline timepoints. Number analyzed signifies participants who were evaluable for this outcome measure at specified timepoints. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
Number analyzed (Participants) | 50 | 52 | 53 | 52
nanograms per milliliter
  Week 1, Day 1: Pre-dose: number analyzed (Participants) | 50 | 52 | 53 | 51
  Week 1, Day 1: Pre-dose | 0.50 (0.0) | 0.50 (0.0) | 0.50 (0.0) | 0.50 (0.0)
  Week 1, Day 1: 1 hour Post-dose: number analyzed (Participants) | 50 | 50 | 52 | 50
  Week 1, Day 1: 1 hour Post-dose | 0.69 (63.7) | 1.85 (247.7) | 2.04 (447.7) | 3.59 (810.5)
  Week 4: Pre-dose: number analyzed (Participants) | 46 | 49 | 50 | 49
  Week 4: Pre-dose | 7.38 (146.8) | 16.22 (246.8) | 55.87 (224.4) | 82.81 (658.3)
  Week 4: 1 hour Post-dose: number analyzed (Participants) | 45 | 47 | 50 | 48
  Week 4: 1 hour Post-dose | 8.45 (140.7) | 21.04 (167.8) | 64.28 (227.6) | 114.95 (322.8)
  Week 4: 4 hours Post-dose: number analyzed (Participants) | 43 | 46 | 48 | 46
  Week 4: 4 hours Post-dose | 12.39 (126.0) | 33.87 (128.3) | 115.04 (191.6) | 222.25 (215.8)
  Week 8: Pre-dose: number analyzed (Participants) | 41 | 47 | 47 | 47
  Week 8: Pre-dose | 7.31 (169.4) | 11.54 (239.7) | 59.94 (193.0) | 103.82 (367.6)
  Week 12: Post-dose: number analyzed (Participants) | 41 | 45 | 47 | 48
  Week 12: Post-dose | 4.66 (182.9) | 13.06 (204.6) | 46.92 (357.1) | 55.51 (1473.5)

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to Week 16
Arm/Group | Placebo | NDI-034858 2 mg | NDI-034858 5 mg | NDI-034858 15 mg | NDI-034858 30 mg
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50 | 0/52 | 0/53 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50 | 0/52 | 1/53 | 0/52
Other Adverse Events (participants affected / at risk) | 9/52 | 16/50 | 10/52 | 16/53 | 15/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | NDI-034858 2 mg (N=50) | NDI-034858 5 mg (N=52) | NDI-034858 15 mg (N=53) | NDI-034858 30 mg (N=52)
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=52) | NDI-034858 2 mg (N=50) | NDI-034858 5 mg (N=52) | NDI-034858 15 mg (N=53) | NDI-034858 30 mg (N=52)
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 3 | 2
Alanine aminotransferase increased (Investigations) | 0 | 3 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 2 | 2 | 2 | 3 | 3
COVID-19 (Infections and infestations) | 1 | 6 | 4 | 6 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 1 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 3 | 2 | 2
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2022-02-04): https://cdn.clinicaltrials.gov/large-docs/39/NCT04999839/Prot_002.pdf
  • Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT04999839/SAP_003.pdf